CLINICAL TRIAL: NCT00568594
Title: A First-in-human, Randomized, Double-blind, Placebo-controlled, Single-ascending Dose (Healthy Volunteers and CHD Patients) and Multiple Dose (CHD Patients) Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of APL180
Brief Title: Safety and Efficacy of APL180 in Healthy Volunteers and Patients With Coronary Heart Disease (CHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CAPL180A2201
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2012-10

CONDITIONS: Coronary Heart Disease
Keywords: Apolipoprotein A-I,; Atherosclerosis,; HDL,; Inflammation,
MeSH Terms: conditions — Coronary Disease; Atherosclerosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: APL180
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APL180
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine: (1) the safety and pharmacokinetics of APL180 administered as a single intravenous infusion in healthy volunteers, and (2) the safety, pharmacokinetics and pharmacodynamics of single and multiple daily intravenous infusions of APL018 in patients with CHD

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteers (ages 18-55 years) and patients with CHD (ages 18 to 75 years) on stable statin therapy for at least 8 weeks, with normal liver and kidney function.
* Women who are post-menopausal, surgically sterile, or practicing effective contraception. Additional birth control details to be provided at screening.
* Body mass index (BMI) must be within the range of 20 to 35 for CHD patients or CHD equivalents.
* Clinical CHD:
* Myocardial infarction (MI), angina, revascularization (e.g. CABG, stent) at least 6 months prior to inclusion
* CHD equivalents:
* symptomatic carotid artery disease (e.g. transient ischemic attack or stroke of carotid origin) or peripheral artery disease or abdominal aortic aneurysm or Diabetes Mellitus (HbA1c ≤9)
* 20% 10 year risk of CHD (Framingham point score: ≥16 (men), ≥23 (women))
* Other clinical forms of atherosclerotic disease including >50 percent stenosis on angiography or ultrasound
* Male subjects, when sexually active, using one form of highly effective contraception (e.g. condom)

Exclusion Criteria for both healthy volunteers and patients:

* Smokers (use of tobacco products in the previous 3 months). Smokers who report cigarette use of more then 10 cigarette per day or have a urinary cotinine level greater then 500 ng/ml.
* Pregnancy.
* Use of any prescription drugs within four (4) weeks prior dosing, or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) within two (2) weeks prior to dosing. Significant illness within two weeks prior to dosing.
* Significant illness within two weeks prior to dosing.
* A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug or any allergic reaction to prior receipt of protein therapies or vaccines.
* Presence of NYHA Class III or IV CHF or unstable angina pectoris.
* MI or within angioplasty (including stenting), acute coronary syndrome (ACS), unstable angina or arterial embolic disease within 6 months prior to dosing.
* Use of certain medications prohibited by the protocol.
* Uncontrolled diabetes (HbA1c > 9).
* Uncontrolled hypertension (Systolic BP >160 mm Hg and/or Diastolic BP >100 mmHg on two consecutive measurements).
* Liver or kidney disease confirmed by abnormal lab values or function.
* Serum creatine kinase CK (CPK) total > 2x.
* CHD equivalent patients with a history of early positive exercise stress test.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, pharmacokinetics and effects on biomarkers of HDL function of APL180 after a single and 7-daily infusions in healthy volunteers (HV) and in patients with coronary heart disease (CHD) | throughout the study

SECONDARY OUTCOMES:
Pharmacokinetic/pharmacodynamic relationship after a single and 7 daily infusions in CHD patients | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigative site
Locations (11):
- Novartis Investigator Site, Philadelphia, Pennsylvania, United States
- Novartis Investigator Site, Antwerp, Belgium
- Novartis Investigator Site, Birkeroed, Denmark
- Israel (3):
  - Novartis Investigator Site, Jerusalem
  - Novartis Investigator Site, Tel Aviv
  - Novartis Investigator Site, Tzrifin
- Novartis Investigator Site, Groningen, Netherlands
- South Africa (3):
  - Novartis Investigator Site, Bloemfontein
  - Novartis Investigator Site, George
  - Novartis Investigator Site, Port Elizabeth
- Novartis Investigator Site, Harrow, United Kingdom

REFERENCES:
- See also: Results for CAPL180A2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3320